CLINICAL TRIAL: NCT03510364
Title: Perceived Social Status as a Determinant of Fat Accretion in Response to Excess Calories: the SSIB Study
Brief Title: Subjective Social Status and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Pennington Biomedical Research Center (Other); University of Florida (Other); University of Alabama at Birmingham (Other); Indiana University (Other)
Responsible Party: Principal Investigator, Emily Dhurandhar, Assistant Professor, Texas Tech University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: IRB2016-571
Record Dates: First submitted 2018-03-12; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Social Dominance; Social Behavior; Eating Behavior
Keywords: Subjective social status; Obesity; High calorie intake; Energy balance; Eating behavior
MeSH Terms: conditions — Obesity; Social Dominance; Social Behavior; Feeding Behavior | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: A prospective feeding study with convenience sampling
Who Masked: Participant
Masking Description: Participants were blinded to the actual study aim. They were told that the aim of the study is to study the relationship between consumption of dietary macronutrient ratios and metabolic rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention (Experimental): All participants consumed a meal that contains 60% of their energy daily energy requirement as a lunch time meal for 14 consecutive days.
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — For the feeding intervention, participants consumed a meal that contains 60% of their energy daily energy requirement as a lunch time meal for 14 consecutive days under observation except during the weekends. To ensure the participant receives 60% of the daily energy requirement as a lunch meal we added a supplemental shake to the standard 1200 kcal meal.

SUMMARY:
Investigators examined the associations between SSS, energy balance, food intake and changes in body composition following a high calorie lunch for 2 weeks.

DETAILED DESCRIPTION:
Subjective social status (SSS) is inversely associated with body fatness. The physiological and psychological effects of low social status may spur increased energy intake as a strategy to buffer against future food scarcity. Investigators' central hypothesis is that females with low SSS will not compensate for excess calorie consumption in a single large meal as well as individuals with high SSS, and will therefore remain in positive energy balance leading to body fat gain in response to daily large meals. Investigators' objective is to understand the influence of SSS on eating behavior, weight gain, and energetic compensation. Investigators conducted a 14-day feeding protocol that consisted of consumption of a lunch-time meal that was 60% of participants' estimated 24-hour energy requirements each day in female participants between 20-50 years, with a body mass index between 25- 30 kg/m2. Free-living food intake was recorded using the Remote Food Photography Method outside of the lab on days 1-2 (early), 7-8 (middle), and 12-13 (late), to measure compensation in response to the large lunch. 24-Hour energy balance, 24 hour intake and post-lunch energy intake were calculated for those days. Investigators measured body composition using Dual energy x ray absorptiometry (DXA), weight and resting energy expenditure at the baseline and at the end of the 14 days of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* between 20-50 years
* body mass index between 25- 30 kg/m2

Exclusion Criteria:

* food allergies or food restrictions
* engaged in any weight reduction program within the past 3 months
* experienced any weight loss or gain of >5% of body weight in the past 6 months for any reason except post-partum weight loss
* taking any medication that suppresses or stimulates appetite
* undergone prior surgical procedures for weight control or liposuction
* current smoker or has not smoked in less than 6 months
* any major diseases including active cancer or cancer requiring treatment in the past 2 years (except non-melanoma skin cancer)
* active or chronic infections (e.g., HIV or TB)
* cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease in the past 6 months
* gastrointestinal disease
* kidney disease
* chronic obstructive airway disease requiring use of oxygen (e.g., emphysema or chronic bronchitis)
* diabetes (type 1 or 2) and taking any anti-diabetic medications and/or controlling the disease via dietary manipulations
* uncontrolled psychiatric disease
* a recent or ongoing problem with drug abuse or addiction
* consume more than three alcoholic drinks per day and has had 7 or more alcoholic beverages in a 24 hour period in the last 12 months
* pregnant or less than 3 months post-partum
* currently nursing or within 6 weeks of having completed nursing
* anticipating a possible pregnancy during the study

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Average 24 hour energy balance (24hr EB) | Six time points ( Days 1, 2, 7, 8, 12 and 13) measured over the two week feeding protocol.
  We measured 24-hr energy balance to assess the association of SSS with positive energy balance in response to a daily large meal perturbation. Twenty four hour energy balance was calculated for each time point as follows, and all six time points were averaged to get an average energy balance over the 2-week period:
  24 hr Energy balance = Average 24 hr Energy intake / Resting Energy Expenditure *1.4 For the early and middle time point 24EB calculations, baseline resting energy expenditure (REE) was used and for late 24hr EB, final REE obtained at the end of the study was used.

SECONDARY OUTCOMES:
Average 24 hour energy intake (24hr EI) over a two week period | Average of six time points ( Days 1, 2, 7, 8, 12 and 13) over a two week period
  Amount of total calories consumed over 24 hours. - consists of breakfast, morning snack, lunch, afternoon snack, dinner, evening snack within 24 hours.
Post-lunch energy intake | Average of six time points (Days 1, 2, 7, 8, 12 and 13) over a two week period
  Amount of total calories consumed after lunch - consists of afternoon snack, dinner, evening snack.
Percent changes in body fat | % change from baseline (day 0) to the end of the intervention period (day 14)
  Changes in the body fat mass
Percent changes in body weight | % change from baseline (day 0) to the end of the intervention period (day 14)
  Changes in the body weight
Changes in adjusted resting energy expenditure | change from baseline (day 0) to the end of the intervention period (day 14)
  Resting energy expenditure (REE) was adjusted to the lean mass. the change in adjusted REE = final adjusted REE - baseline adjusted REE

IPD SHARING:
Plan to Share IPD: No